CLINICAL TRIAL: NCT04081324
Title: Safety, Tolerability, and Pharmacokinetics of Lasmiditan in Healthy Chinese Subjects
Brief Title: A Study of Lasmiditan in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17022; H8H-MC-LAIC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo administered orally on Day 1 and repeated doses on Days 4 to 10 (7 days of dosing).
  Interventions: Drug: Placebo
- 50 milligram (mg) Lasmiditan (Experimental): Participants received 50 mg lasmiditan administered orally once on the morning of Day 1 after an overnight fast of at least 8 hours. Following a period of at least 72 hours without dosing, participants received multiple once-daily oral doses of 50 mg lasmiditan on Days 4 to 10 (7 days of dosing) after overnight fasts of at least 8 hours prior to each dose.
  Interventions: Drug: Lasmiditan
- 100 mg Lasmiditan (Experimental): Participants received 100 mg lasmiditan administered orally once on the morning of Day 1 after an overnight fast of at least 8 hours. Following a period of at least 72 hours without dosing, participants received multiple once-daily oral doses of 100 mg lasmiditan on Days 4 to 10 (7 days of dosing) after overnight fasts of at least 8 hours prior to each dose.
  Interventions: Drug: Lasmiditan
- 200 mg Lasmiditan (Experimental): Participants received 200 mg lasmiditan administered orally once on the morning of Day 1 after an overnight fast of at least 8 hours. Following a period of at least 72 hours without dosing, participants received multiple once-daily oral doses of 200 mg lasmiditan on Days 4 to 10 (7 days of dosing) after overnight fasts of at least 8 hours prior to each dose.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: 100 mg Lasmiditan; 200 mg Lasmiditan; 50 milligram (mg) Lasmiditan
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This is a study of lasmiditan in healthy Chinese participants. The purposes are:

* To evaluate the safety of lasmiditan
* To learn more about how the body processes lasmiditan

The study will last up to 50 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy Chinese (all 4 biological grandparents and both biological parents to be of Chinese origin) males or females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.0 to 32.0 kilograms per square meter, inclusive
* Are able and willing to give signed informed consent

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds or any components of the formulation
* Have an abnormal blood pressure and/or pulse rate as determined clinically significant by the investigator
* Have a history of, show evidence of, or are undergoing treatment for significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* Have a history of central nervous system (CNS) conditions such as strokes, transient ischemic attack, significant head trauma, CNS infections, migraines, brain surgery, or any other neurological conditions that, in the opinion of the investigator, increases the risk of participating in the study
* Regularly use known drugs of abuse and/or show positive findings on drug screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 50 Milligram (mg) Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Started | 6 | 10 | 10 | 10
Received At Least One Dose of Study Drug | 6 | 10 | 10 | 10
Completed | 6 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 50 mg Lasmiditan: Participants received 50 mg lasmiditan administered orally once on the morning of Day 1 after an overnight fast of at least 8 hours. Following a period of at least 72 hours without dosing, participants received multiple once-daily oral doses of 50 mg lasmiditan on Days 4 to 10 (7 days of dosing) after overnight fasts of at least 8 hours prior to each dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | Total
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.20 (9.75) | 31.90 (5.82) | 33.40 (4.88) | 30.00 (5.66) | 31.70 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 3 | 9
  Male | 4 | 7 | 9 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 10 | 10 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 10 | 10 | 10 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 6 | 10 | 10 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity AUC(0-∞) of Lasmiditan
Description: PK: Area Under the Concentration Versus Time Curve from time zero to infinity AUC(0-∞) of Lasmiditan after single dose (Day 1).
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 10 | 10 | 10
nanogram*hour per milliliter (ng*h/mL) | 385 (48) | 829 (34) | 1990 (34)

2. Primary Outcome: PK: Area Under the Plasma Concentration-Time Curve Over a 24-Hour Dosing Interval (AUCτ) of of Lasmiditan
Description: PK: AUCτ of of Lasmiditan was calculated based on the of Lasmiditan plasma concentration time curve from time 0 hour (hr) to time 24 hr (tau [τ]) when Lasmiditan was administered after single dose (day 1) and multiple doses (Day 10).
Time Frame: Day 1 (Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, and 24 hours post-dose) and Day 10 (Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose)
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 10 | 10 | 10
ng*h/mL
  Day 1 | 378 (47) | 809 (34) | 1950 (34)
  Day 10 | 429 (36) | 898 (28) | 2140 (33)

3. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Lasmiditan
Description: PK: Maximum Observed Drug Concentration (Cmax) of Lasmiditan after single dose (day 1) and multiple doses (Day 10).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 10 | 10 | 10
nanograms per milliliter (ng/mL)
  Day 1 | 69.6 (48) | 154 (37) | 359 (33)
  Day 10 | 78.8 (50) | 187 (28) | 394 (37)

4. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Lasmiditan
Description: PK: Time to Maximum Observed Plasma Concentration (tmax) of Lasmiditan after single dose (Day 1) and multiple doses (Day 10).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 10 | 10 | 10
hours (h)
  Day 1 | 1.50 [0.50 to 2.50] | 1.50 [0.50 to 2.50] | 1.50 [1.00 to 2.97]
  Day 10 | 1.75 [0.50 to 2.50] | 1.50 [1.00 to 2.00] | 1.50 [0.50 to 2.50]

ADVERSE EVENTS:
Time Frame: Baseline, Up to 4 months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/6 | 9/10 | 10/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 50 mg Lasmiditan (N=10) | 100 mg Lasmiditan (N=10) | 200 mg Lasmiditan (N=10)
Atrioventricular block first degree (Cardiac disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 5 (6) | 5 (10) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 3 (11) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Puncture site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (4) | 6 (10) | 6 (16) | 2 (2)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil percentage increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary casts (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (11) | 5 (13) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 3 (7) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 9 (29) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04081324/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04081324/SAP_001.pdf